CLINICAL TRIAL: NCT05697250
Title: High Versus Low Power Settings During Ureteroscopic Laser Lithotripsy - a Prospective, Randomised Clinical Trial
Brief Title: High Versus Low Power Settings During Ureteroscopic Laser Lithotripsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550740
Record Dates: First submitted 2022-12-29; First posted 2023-01-25 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: The patients are randomised to ureteroscopic stone treatment with Thulium Fiber Laser with either low or high laser settings. The ureteroscopic procedures are performed in a standardised manner irrespective of the laser settings, and follow-up is similar in both groups.
Who Masked: Outcomes Assessor
Masking Description: Stone free status is assessed on low dose CT 3 months post endoscopically by an outcome assessor blinded to the randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - low power laser settings (Experimental): 4-6 Watts, short pulse mode. 0.4 - 0.6 J at 10 Hz.
  Interventions: Other: Laser power settings (Thulium Fiber Laser)
- Group 2 - high power laser settings (Experimental): 16-18 Watts, short pulse mode. 0.4 J / 40 Hz, 0.6 J / 30 Hz or 0.8 J / 20 Hz.
  Interventions: Other: Laser power settings (Thulium Fiber Laser)

INTERVENTIONS:
Other: Laser power settings (Thulium Fiber Laser) — Ureteroscopic lithotripsy using low power laser settings (0.4 - 0.6 J at 10 Hz corresponding to 2.4 - 6.0 Watts) or high power laser settings (0.4 J at 40 Hz, 0.6 J at 30 Hz or 0.8 J at 20 Hz corresponding to 16 - 18 Watts).

SUMMARY:
The primary aim of the study is to compare the operative times following ureteroscopic lithotripsy for renal stones with Thulium Fiber Laser using low and high power settings.

Secondary aims are to compare the results of low and high power settings in terms of stone free rates, laser time, laser activation patterns, intraoperative and postoperative complications.

Patients ≥ 18 years with renal stones (8-25 mm) scheduled for ureteroscopic lithotripsy at the Day Surgery Clinic at Haukeland University Hospital in Bergen, Norway, are eligible for inclusion in the study. After written consent and inclusion, patients are randomised to laser lithotripsy using either low power settings (Group 1: 4-6 Watt, short pulse mode) or high power settings (Group 2: 16-18 Watt, short pulse mode). The ureteroscopic procedures are performed in general anaesthesia using a standardised technique. All patients are followed up with a low dose CT scan 3 months post endoscopically to assess stone free status as well as a consultation at the outpatient clinic.

Results and data for the two randomisation groups are compared according to the aims of the study.

DETAILED DESCRIPTION:
BACKGROUND: The Holmium:Yttrium-Aluminium-Garnet (Ho:YAG) has been considered the gold-standard laser for ureteroscopy (URS) because of its versatility, with the ability to break all kinds of stones in the urinary tract as well as tumor- and soft tissue ablation. Recently, a new Thulium fiber laser (TFL) has been introduced, with more favourable basic physical characteristics. Previous pre-clinical studies have predicted TFL lithotripsy to be up to four times faster than Ho:YAG lithotripsy using the same power settings. Earlier this year the present investigators published the first clinical randomised trial comparing the outcomes after ureteroscopic lithotripsy using TFL and Ho:YAG. The study demonstrated that the TFL gained superior stone free rate (SFR) compared to Ho:YAG, in addition to lower complication rate and shorter operative times. Due to the study, the investigators believe the TFL is emerging as the laser of choice. In the study very low laser settings were shown to be highly efficient using TFL during URS lithotripsy. However, no consensus exists on the preferred laser settings for the TFL during this procedure, and a variety of different settings have been suggested included high power settings as high as 45 Watts (W).

To date, there are no clinical randomised trials comparing different laser settings for TFL to determine what is optimal regarding the clinical outcomes.

AIMS OF THE STUDY: The primary aim of the study is to compare the operative times following URS lithotripsy for renal stones with TFL using low and high power settings. Secondary aims are to compare the results of low and high power settings in terms of SFR, laser time, laser activation patterns, intraoperative and postoperative complications.

STUDY DESIGN: The study is planned as a prospective randomized trial. All patients ≥ 18 years scheduled to URS lithotripsy for renal stones, 8-25 mm, at the day surgery unit at Haukeland University Hospital (HUH) are invited to be enrolled in the study. After written informed consent, patients are randomized to URS TFL lithotripsy with either low or high power laser settings.

LASER SETTINGS: The laser settings in the two study groups are standardized and need to be maintained throughout the procedure.

Group 1 - low power (4-6W), short pulse: 0.4 - 0.6 Joules (J) at 10 Herz (Hz) Group 2 - high power (16-18W), short pulse: 0.4 J / 40 Hz 0.6 J / 30 Hz 0.8 J / 20 Hz

Standard start-up settings in Group 1 (low power) is 0.4J / 10Hz (4W) and in Group 2 (high power) 0.4J / 40Hz (16W).

THE URS PROCEDURE: The URS procedure is performed in general anaesthesia and prophylactic antibiotics prior to surgery start will be administered according to the department's guidelines, either according to urine culture or current local regime.

The procedure starts with a cystoscopy followed by semirigid URS when considered appropriate. A safety guide wire and an access sheath can be used at the surgeon's discretion but is routinely omitted during URS at HUH. Balloon dilatation is performed on demand. Both semirigid and flexible ureteroscopes can be used for the endoscopy. Room-tempered, gravitational irrigation fluid at 60 cm height is used throughout the procedure. When reaching the stone, the envelope revealing the result of randomization for either high or low laser settings is opened. A 150μm laser fiber can be used for stone disintegration. The stone is disintegrated using TFL with predefined settings as described below and according to the randomization group. To make the procedures as similar as possible, the stone should be dusted/disintegrated to as small particles as possible rather than fragmented and retrieved. Only residual particles not suitable for further disintegration can be retrieved at the end of the procedure to render the patient stone free.

A double J-stent can be placed after the procedure if deemed necessary, and if so, this is removed according to standard routine after 1-2 weeks in the outpatient clinic.

FOLLOW-UP: Follow-up with computed tomography (CT) is performed at 3 months post endoscopically for all patients to assess stone free status and exclude a ureteral stricture in addition to a clinical consultation.

ETHICAL CONSIDERATIONS AND APPROVALS: All patients eligible for inclusion in the study will receive oral and written information. Participation in the study is voluntarily, and the patient can choose to withdraw at any point during the study process. Inclusion in the study will only be done after the consent form is signed.

The study is approved by The National Committees for Research Ethics in Norway (REK: 550740). In addition, application for approval by The Data Protection Authorities at Haukeland University Hospital has been sent.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years scheduled for URS lithotripsy for renal stones, 8-25 mm, at the day surgery unit at Haukeland University Hospital

Exclusion Criteria:

* Concomitant ureteral stone
* Urinary diversion
* Active infection
* Untreated cancer in the upper urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Operative time | During surgery (approximately 1 hour), registered immediately after surgery
  Surgical time in minutes, counted from start of the procedure with insertion of the cystoscope until emptying the bladder in the end.

SECONDARY OUTCOMES:
Stone free rate | 3 months post endoscopically
  Assessment of stone free status (or the presence of residual fragments) on low dose CT 3 months post endoscopically.
Laser activation patterns - duration | During surgery (approximately 1 hour), registered immediately after surgery
  Duration of laser activation periods during laser lithotripsy in seconds
Laser activation patterns - number | During surgery (approximately 1 hour), registered immediately after surgery
  Number of laser activation periods during laser lithotripsy
Intraoperative complications | During surgery (approximately 1 hour), registered immediately after surgery
  Complications occurred during the endoscopic procedure (bleeding, perforation, avulsion, mucosal abrasion, blurred vision)
Post operative complications | After surgery until 3 months post endoscopically.
  Complications occurred after the endoscopic procedure (up to 3 months post endoscopically).

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ulvik, Assoc Prof, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No